CLINICAL TRIAL: NCT04847336
Title: IMAGINE EURO (Improving MAternal Newborn carE In the EURO Region): Maternal and Newborn Health Service Preparedness, Quality and Resilience, Among Countries of the WHO European Region, During the COVID-19 Pandemic
Brief Title: Improving MAternal Newborn carE In the in the WHO European Region During COVID-19 Pandemic
Acronym: IMAgiNE-EURO
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: WHO Collaborating Centre for Maternal and Child Health, Trieste (Other)
Collaborators: IRCCS Burlo Garofolo (Other); NGO Babysteps (Unknown); Roda - Parents in Action (Unknown); INED - Institut National d'Etudes Démographiques (Unknown); School of Public Health, Bielefeld University (Unknown); Riga Stradins University (Other); BLL-Beruffsverband vun den Laktationsberoderinnen zu Lëtzebuerg asbl (Unknown); UiT The Arctic University of Norway (Other); Childbirth with Dignity Foundation (Unknown); Instituto de Saude Publica da Universidade do Porto (Other); Administraçao Regional de Saude do Algarve - ACES Central - URAP - Albufeira (Unknown); Associação Portuguesa pelos Direitos da Mulher na Gravidez e Parto (Unknown); Universidade Europeia, Lisbon (Unknown); SAMAS Association (Unknown); Centar za mame (Unknown); National Institute of Public Health, Slovenia (Other Government); Medical Anthropology Research Center (MARC, URV) (Unknown); Göteborg University (Other); University of Exeter (Other)
Responsible Party: Principal Investigator, Marzia Lazzerini, paediatrician, DTMH, Msc, PhD Director SS WHO Collaborating Center IRCCS Burlo Trieste Italy, WHO Collaborating Centre for Maternal and Child Health, Trieste
Other Study IDs: IRB-BURLO 05/2020
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Quality of Care During Childbirth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women: Women of any age who gave births in hospitals from WHO European Region, from 1 march 2020
  Interventions: Other: No intervention is planned
- Health workers: Health workers directly involved in assistance at childbirth (pregnancy, childbirth and peripartum) at hospital level in WHO European Region, from 1 march 2020
  Interventions: Other: No intervention is planned

INTERVENTIONS:
Other: No intervention is planned — No intervention is planned

SUMMARY:
BACKGROUND COVID-19 response is heavily impacting the availability of essential health services, especially services for pregnant women and newborns that cannot be delayed or rapidly reorganized in other settings. In the current pandemic, due to multiple factors access to high quality and timely maternal and newborn (MN) health care is threatened. Major concerns have also been raised with respect to maternal rights and on disruption of essential practices and increased medicalization of care, despite existing WHO guidance.

Based on preliminary reports heterogeneities in practices is expected within the WHO European Region, with major inequities (eg women experiencing disruption of essential MC health services only in selected countries or areas within the countries, while having access to adequate care in others).

With IMAgiNE EURO we aim at conducting a survey to explore the health service preparedness, quality and resilience, with a specific focus on health services around the time of childbirth, in the WHO European Region during COVID-19 pandemic, and to make available data, which, in collaboration with WHO and other partners, can contribute in improving the quality of MN health care.

HYPHOTESIS AND SIGNIFICANCE

* This project has been developed in coordination with WHO Regional Office for Europe (EURO) and other partners, and ultimately aims at making available and disseminate data that can help improving the quality of MN health services in the Region. Collecting data on the quality of essential MN health services across different countries within the WHO European Region will help addressing specific gaps and planning coordinate response to improve quality of MN care and improve MN health outcomes.
* The project will also offer the opportunity to develop tools and methods to monitor the quality of MN health care across different countries and settings.
* The project will establish and consolidate a research network

Primary objective:

1. Record, analyse, and describe data on MN health service preparedness, quality and resilience - with a specific focus around the time of childbirth as measured both from health workers and women perspectives- across different countries within the WHO European Region, during COVID-19 pandemic.

Secondary objectives: 2.Develop tools and methods to measure, through rapid online surveys, the quality of MN health care across different countries and settings 3.Establish and consolidate a research network

ELIGIBILITY:
Inclusion Criteria:

1. Women of any age who gave births in hospitals, from 1 march 2020
2. Health workers directly involved in assistance at childbirth (pregnancy, childbirth and peripartum) at hospital level, from 1 march 2020

Exclusion Criteria:

1. For women: refusal to participate; home births
2. For health workers: personnel not directly involved in the routine care t childbirth (es physiotherapist, philologist), refusal to participate; absence from work for more than 2 months out of the 4 months immediately before the survey; less than 1 year of experience

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be collected among mothers and among health workers providing care to mothers or infants.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Maternal and Newborn Care Index - mean | March 2020 to March 2021
  variable from 0 to 100 points

SECONDARY OUTCOMES:
Quality of Maternal and Newborn Care Index - total value | March 2020 to March 2021
  variable from 0 to 400 points
Index of Quality of Maternal and Newborn Care - value by domains | March 2020 to March 2021
  * Index for availability of human and physical resources (variable from 0 to 100 points)
  * Index for provision of care (variable from 0 to 100 points)
  * Index for experience of care (variable from 0 to 100 points)
  * Index for COVID-19 related care (variable from 0 to 100 points)
Frequency of specific indicators/quality measure | March 2020 to March 2021
  * Caesarean section rate
  * Episiotomy rate
  * Availability of specific resources

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Lazzerini, PhD Dr, Principal Investigator — WHO Collaborating Center for Maternal and Child Health - IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazzerini M, Valente EP, Covi B, Semenzato C, Ciuch M. Use of WHO standards to improve quality of maternal and newborn hospital care: a study collecting both mothers' and staff perspective in a tertiary care hospital in Italy. BMJ Open Qual. 2019 Feb 13;8(1):e000525. doi: 10.1136/bmjoq-2018-000525. eCollection 2019. PMID 30997420
- [Background] Lazzerini M, Mariani I, Semenzato C, Valente EP. Association between maternal satisfaction and other indicators of quality of care at childbirth: a cross-sectional study based on the WHO standards. BMJ Open. 2020 Sep 14;10(9):e037063. doi: 10.1136/bmjopen-2020-037063. PMID 32928854
- [Background] Lazzerini M, Semenzato C, Kaur J, Covi B, Argentini G. Women's suggestions on how to improve the quality of maternal and newborn hospital care: a qualitative study in Italy using the WHO standards as framework for the analysis. BMC Pregnancy Childbirth. 2020 Apr 6;20(1):200. doi: 10.1186/s12884-020-02893-0. PMID 32252686
- [Derived] Galle A, Berghman H, D'Hauwers S, Vaerewijck N, Valente EP, Mariani I, Bomben A, Delle Vedove S, Lazzerini M; IMAgiNE EURO Study Group. Quality of care at childbirth during the COVID-19 pandemic in Belgium: a cross-sectional study based on WHO standards. BMJ Open. 2024 Dec 27;14(12):e086937. doi: 10.1136/bmjopen-2024-086937. PMID 39732493
- [Derived] Zaigham M, Linden K, Elden H, Delle Vedove S, Mariani I, Kongslien S, Drandic D, Pumpure E, Drglin Z, Costa R, Sarantaki A, de Labrusse C, Miani C, Otelea MR, Liepinaitiene A, Baranowska B, Rozee V, Valente EP, Vik ES, Kurbanovic M, Jakovicka D, Bohinec A, Dias H, Metallinou D, Mueller AN, Batram-Zantvoort S, Handra CM, Mizgaitiene M, Tataj-Puzyna U, Bomben A, Nedberg IH, Voitehovica E, Pinto TM, Lykeridou A, Grylka-Baeschlin S, Jazdauskiene S, Szlendak B, Sacks E, Lazzerini M; IMAgiNE EURO Study group. Trends in the quality of maternal and neonatal care in Sweden and Norway as compared to 12 WHO European countries: A cross-sectional survey investigating maternal perspectives during the COVID-19 pandemic. Acta Obstet Gynecol Scand. 2024 Dec;103(12):2485-2498. doi: 10.1111/aogs.14994. Epub 2024 Oct 21. PMID 39431577
- [Derived] Grylka-Baeschlin S, Gemperle M, Mariani I, Abderhalden-Zellweger A, Miani C, Zenzmaier C, Mueller AN, Batram-Zantvoort S, Koenig-Bachmann M, De Labrusse C, Arendt M, Vedove SD, Pfund A, Simon I, Valente EP, Lazzerini M; IMAgiNE Euro Study Group. Women 's perception on the quality of maternal and newborn care during the COVID-19 pandemic in German-speaking countries: Findings from the IMAgiNE EURO project comparing data from Germany, Switzerland and Austria. Midwifery. 2025 Jan;140:104209. doi: 10.1016/j.midw.2024.104209. Epub 2024 Oct 11. PMID 39423767
- [Derived] Valente EP, Mariani I, Bomben A, Morano S, Gemperle M, Otelea MR, Miani C, Elden H, Sarantaki A, Costa R, Baranowska B, Konig-Bachmann M, Kongslien S, Drandic D, Rozee V, Nespoli A, Abderhalden-Zellweger A, Nanu I, Batram-Zantvoort S, Linden K, Metallinou D, Dias H, Tataj-Puzyna U, D'Costa E, Nedberg IH, Kurbanovic M, de La Rochebrochard E, Fumagalli S, Grylka-Baeschlin S, Handra CM, Zaigham M, Orovou E, Barata C, Szlendak B, Zenzmaier C, Vik ES, Liepinaitiene A, Drglin Z, Arendt M, Sacks E, Lazzerini M; Improving MAternal Newborn carE in the EURO Region (IMAgiNE EURO) Study Group. Health workers' perspectives on the quality of maternal and newborn health care around the time of childbirth: Results of the Improving MAternal Newborn carE in the EURO Region (IMAgiNE EURO) project in 12 countries of the World Health Organization European Region. J Glob Health. 2024 Sep 6;14:04164. doi: 10.7189/jogh.14.04164. PMID 39238363
- [Derived] Artzi-Medvedik R, Mariani I, Valente EP, Lazzerini M, Chertok IA. Factors associated with exclusive breastfeeding in Israel during the COVID-19 pandemic: a subset of the IMAgiNE EURO cross-sectional study. Int Breastfeed J. 2023 Jun 9;18(1):30. doi: 10.1186/s13006-023-00568-y. PMID 37296409
- [Derived] Geremia S, Valente EP, Mariani I, Dalena P, Lazzerini M. Women's suggestions on how to improve the quality of maternal and newborn care during the COVID-19 pandemic in Italy: A co-occurrence network analysis. J Glob Health. 2023 May 5;13:06013. doi: 10.7189/jogh.13.06013. PMID 37144478
- [Derived] Pumpure E, Jakovicka D, Mariani I, Vaska A, Covi B, Valente EP, Jansone-Santare G, Knoka AR, Vilcane KP, Rezeberga D, Lazzerini M; IMAgiNE EURO study group. Women's perspectives on the quality of maternal and newborn care in childbirth during the COVID-19 pandemic in Latvia: Results from the IMAgiNE EURO study on 40 WHO standards-based quality measures. Int J Gynaecol Obstet. 2022 Dec;159 Suppl 1(Suppl 1):97-112. doi: 10.1002/ijgo.14461. PMID 36530013
- [Derived] Otelea MR, Simionescu AA, Mariani I, Valente EP, Nanu MI, Nanu I, Handra CM, Covi B, Lazzerini M; IMAgiNE EURO Study Group. Women's assessment of the quality of hospital-based perinatal care by mode of birth in Romania during the COVID-19 pandemic: Results from the IMAgiNE EURO study. Int J Gynaecol Obstet. 2022 Dec;159 Suppl 1(Suppl 1):126-136. doi: 10.1002/ijgo.14482. PMID 36530009
- [Derived] Lazzerini M, Valente EP, Covi B, Rozee V, Costa R, Otelea MR, Abderhalden-Zellweger A, Wegrzynowska M, Linden K, Arendt M, Brigidi S, Miani C, Pumpure E, Radetic J, Drandic D, Cerimagic A, Nedberg IH, Liepinaitiene A, Rodrigues C, de Labrusse C, Baranowska B, Zaigham M, Castaneda LM, Batram-Zantvoort S, Jakovicka D, Ruzicic J, Juciute S, Santos T, Gemperle M, Tataj-Puzyna U, Elden H, Mizgaitiene M, Lincetto O, Sacks E, Mariani I; IMAgiNE EURO study group. Rates of instrumental vaginal birth and cesarean and quality of maternal and newborn health care in private versus public facilities: Results of the IMAgiNE EURO study in 16 countries. Int J Gynaecol Obstet. 2022 Dec;159 Suppl 1(Suppl 1):22-38. doi: 10.1002/ijgo.14458. PMID 36530007
- [Derived] Drandic D, Drglin Z, Mihevc Ponikvar B, Bohinec A, Cerimagic A, Radetic J, Ruzicic J, Kurbanovic M, Covi B, Valente EP, Mariani I, Lazzerini M; IMAgiNE EURO study group. Women's perspectives on the quality of hospital maternal and newborn care around the time of childbirth during the COVID-19 pandemic: Results from the IMAgiNE EURO study in Slovenia, Croatia, Serbia, and Bosnia-Herzegovina. Int J Gynaecol Obstet. 2022 Dec;159 Suppl 1(Suppl 1):54-69. doi: 10.1002/ijgo.14457. PMID 36530003
- [Derived] Chertok IA, Artzi-Medvedik R, Arendt M, Sacks E, Otelea MR, Rodrigues C, Costa R, Linden K, Zaigham M, Elden H, Drandic D, Grylka-Baeschlin S, Miani C, Valente EP, Covi B, Lazzerini M, Mariani I. Factors associated with exclusive breastfeeding at discharge during the COVID-19 pandemic in 17 WHO European Region countries. Int Breastfeed J. 2022 Dec 2;17(1):83. doi: 10.1186/s13006-022-00517-1. PMID 36461061
- [Derived] Valente EP, Covi B, Mariani I, Morano S, Otalea M, Nanu I, Nanu MI, Elden H, Linden K, Zaigham M, Vik ES, Kongslien S, Nedberg I, Costa R, Rodrigues C, Dias H, Drandic D, Kurbanovic M, Sacks E, Muzigaba M, Lincetto O, Lazzerini M; IMAgiNE EURO Study Group. WHO Standards-based questionnaire to measure health workers' perspective on the quality of care around the time of childbirth in the WHO European region: development and mixed-methods validation in six countries. BMJ Open. 2022 Apr 8;12(4):e056753. doi: 10.1136/bmjopen-2021-056753. PMID 35396296
- [Derived] Lazzerini M, Covi B, Mariani I, Drglin Z, Arendt M, Nedberg IH, Elden H, Costa R, Drandic D, Radetic J, Otelea MR, Miani C, Brigidi S, Rozee V, Ponikvar BM, Tasch B, Kongslien S, Linden K, Barata C, Kurbanovic M, Ruzicic J, Batram-Zantvoort S, Castaneda LM, Rochebrochard E, Bohinec A, Vik ES, Zaigham M, Santos T, Wandschneider L, Viver AC, Cerimagic A, Sacks E, Valente EP; IMAgiNE EURO study group. Quality of facility-based maternal and newborn care around the time of childbirth during the COVID-19 pandemic: online survey investigating maternal perspectives in 12 countries of the WHO European Region. Lancet Reg Health Eur. 2022 Feb;13:100268. doi: 10.1016/j.lanepe.2021.100268. Epub 2021 Dec 24. PMID 34977838
- See also: Webpage were survey links for women (in more than 20 languages) and health workers (in more than 10 languages)are available. — http://www.burlo.trieste.it/ricerca/imagine-euro-improving-maternal-newborn-care-euro-region